CLINICAL TRIAL: NCT04276415
Title: Phase 1, Multicenter, Open-Label, First-in-Human Study of DS-6157a in Subjects With Advanced Gastrointestinal Stromal Tumor
Brief Title: DS-6157a in Participants With Advanced Gastrointestinal Stromal Tumor (GIST)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a business decision.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS6157-A-U101
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal stromal tumors; DS-6157a; Anti-drug antibody conjugate; G-protein coupled receptor 20 (GPR20)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: DS-6157a (Experimental): Participants with advanced gastrointestinal stromal tumor (GIST) who will receive an intravenous infusion of DS-6157a (escalating doses starting at 1.6 mg/kg).
  Interventions: Drug: DS-6157a
- Dose Expansion: Cohort 1 (3rd line or later) treated at RDE (Experimental): Participants with advanced gastrointestinal stromal tumor (GIST) who have progressed on or are intolerant to imatinib (IM) and at least one post-IM treatment will receive DS-6157a at the recommended dose for expansion (RDE) based on the Dose Escalation phase.
  Interventions: Drug: DS-6157a
- Dose Expansion: Cohort 2 (2nd line) treated at RDE (Experimental): Participants with advanced gastrointestinal stromal tumor (GIST) who have progressed on imatinib (IM) and had not received a post-IM treatment (2nd line) will receive DS-6157a at the recommended dose for expansion (RDE) based on the Dose Escalation phase.
  Interventions: Drug: DS-6157a

INTERVENTIONS:
Drug: DS-6157a — Administered as a single agent intravenously (IV) every 3 weeks

SUMMARY:
This study will assess the safety, efficacy, and pharmacokinetics of DS-6157a in participants with advanced gastrointestinal stromal tumors (GIST).

DETAILED DESCRIPTION:
This study is a two-part, multicenter, open-label, multiple-dose, first-in-human study of the antibody-drug conjugate (ADC) DS-6157a given as a single agent to participants with gastrointestinal stromal tumor (GIST).

This study will include 2 parts:

1. Dose Escalation (Part 1)
2. Dose Expansion (Part 2)

Dose Escalation: Participants with histopathologically documented advanced GIST not amenable to curative therapy may be included in which the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of DS-6157a monotherapy will be determined.

Dose Expansion: Once the RDE(s) is established for DS-6157a (Part 1), enrollment in Dose Expansion (Part 2) will commence in 2 cohorts. Participants with GIST who have progressed on or are intolerant to imatinib (IM) and at least one post-IM treatment will be enrolled in Cohort 1, and participants with GIST who progressed on IM and had not received a post-IM treatment (2nd line) will be enrolled in Cohort 2.

The study was terminated after Dose Escalation and the study never proceeded to the Dose Expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least 20 years old in Japan or 18 years old in other countries at the time of signature of the informed consent form (ICF), following local regulatory requirements
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Has histopathologically documented unresectable and/or metastatic GIST meeting the criteria below:
* Dose Escalation (Part 1): Participants should meet one of the following criteria:

  1. (For US sites only) Participants with GIST who have progressed on or are intolerant to imatinib (IM) and at least one post-IM treatment or who are not candidates for post-IM standard of care treatment
  2. (For Japan sites only) Participants with GIST who have received all the existing standard of care treatments or who are not candidates for one or more available post-IM standard of care treatments
  3. Participants with GIST who are not candidates for IM or curative intent surgical treatment (i.e., participants without activating KIT or platelet-derived growth factor receptor alpha (PDGFRa) mutations, with PDGFRa D842V mutations, or are KIT negative by local results)
* Dose Expansion (Part 2) Cohort 1: Participants with GIST who have progressed on or are intolerant to IM and at least one post-IM treatment
* Dose Expansion (Part 2) Cohort 2: Participants with GIST who have progressed on IM and had not received a post-IM treatment (2nd line)
* Consents to provide fresh tumor biopsy tissue samples both before and on DS-6157a treatment for the measurement of GPR20 levels by immunohistochemistry and other biomarkers
* Has a left ventricular ejection fraction (LVEF) ≥50% by either echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) within 28 days before study treatment
* Has at least 1 measurable lesion based on RECIST Version 1.1 as assessed by the Investigator
* Has adequate organ function within 7 days before the start of study treatment, defined as:

  1. Platelet count ≥100,000/mm^3
  2. Hemoglobin ≥8.5 g/dL
  3. Absolute neutrophil count ≥1,500/mm^3
  4. Creatinine clearance ≥50 mL/min
  5. Aspartate aminotransferase ≤3 × upper limit of normal (ULN) (if liver metastases are present, ≤5 × ULN)
  6. Alanine aminotransferase ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  7. Total bilirubin ≤1.5 × ULN or ≤3.0 × ULN for participants with documented history of Gilbert's Syndrome
* Has an adequate treatment washout period prior to start of study treatment, defined as:

  1. Major surgery: ≥4 weeks (or 2 weeks for minor surgeries)
  2. Radiation therapy: ≥3 weeks (or 2 weeks for palliative radiation excluding pelvic radiation)
  3. Systemic anti-cancer therapy (except for anti-androgen for prostate cancer and bisphosphonate, denosumab, or medroxyprogesterone acetate for bone metastases):

     * Cytotoxic chemotherapy: ≥3 weeks or 5 times the terminal elimination half-life (t½) of the chemotherapeutic agent, whichever is shorter
     * Antibody and antibody-conjugates therapy: ≥3 weeks or 5 times the t½, whichever is longer
     * Prior tyrosine kinase inhibitors (TKIs): washout period from 2 to 21 days depending on the TKI
     * Immunotherapy: ≥4 weeks.
* Male participants with female partners of childbearing potential and female participants of child-bearing potential must agree to use a highly effective form of contraception, or avoid intercourse during and upon completion of the study and for at least 4 months (for males) and for at least 7 months (for females) after the last dose of study drug.

Exclusion Criteria:

* History of an allogeneic bone marrow or solid organ transplant within 3 months before the start of study treatment
* Concomitant treatment with any medication that is classified as having a known risk of Torsades de pointes should be avoided from the start of study treatment through the end of Cycle 3
* Prophylactic administration of granulocyte colony-stimulating factor (G-CSF), filgrastim, pegfilgrastim, erythropoietin, or the transfusion of blood, red blood cells, or platelets within 14 days before the start of treatment and during Cycle 1. Chronic therapy with erythropoietin at stable dose that started at least 14 days before the first dose of DS-6157a may continue.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, Grade ≤1. Participants with chronic Grade 2 toxicities may be eligible.
* Has spinal cord compression or clinically active central nervous system (CNS) metastases (including brain metastases), defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms
* Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product
* Has a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety, efficacy, or any other assessments of the investigational regimen
* Has a documented history of myocardial infarction or unstable angina within 6 months before study treatment
* Has a medical history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or a serious cardiac arrhythmia requiring treatment
* Has a corrected QT by Fridericia's formula (QTcF), of >470 ms based on the average of triplicate 12-lead electrocardiogram (ECG) per local read
* Has a documented history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Has clinically significant pulmonary compromise or requirement for supplemental oxygen
* Has clinically significant corneal disease
* Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Has active human immunodeficiency virus (HIV) infection as determined by plasma HIV RNA viral load.
* Has evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, as manifest by the detectable viral load (HBV-DNA or HCV-RNA, respectively)
* Is a lactating mother (women who are willing to temporarily interrupt breastfeeding will also be excluded), or pregnant as confirmed by pregnancy tests performed within 7 days before study treatment
* Women who plan to become pregnant while in the study and for at least 7 months after the last administration of study treatment
* Men who plan to father a child while in the study and for at least 4 months after the last administration of study treatment
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, substance abuse, or other medical condition that would increase the risk of toxicity or interfere with participation of the participant or evaluation of the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (5):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University of St. Louis, St Louis, Missouri
  - Oregon Health and Science University, Portland, Oregon
  - MD Anderson, Houston, Texas
- National Cancer Center Hospital East, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants who met all inclusion and no exclusion criteria were enrolled and received treatment at 5 clinic sites in the United States and Japan.
Pre-assignment Details: Dose Escalation (Part 1) was designed to establish the maximum tolerated dose and recommended dose of expansion (RDE) for DS-6157a. Dose-Expansion (Part 2) was expected to start at the RDE to further characterize the safety and tolerability, pharmacokinetics profile, and efficacy of DS-6157a; however, due to lower than anticipated efficacy in Part 1, the Sponsor decided to terminate the study prior to Dose Expansion. Efficacy analyses were limited in Part 1; no analyses in Part 2 were conducted.
Groups:
- Dose Escalation: DS-6157a 1.6 mg/kg: Participants with advanced gastrointestinal stromal tumor (GIST) who received an intravenous (IV) infusion of DS-6157a 1.6 mg/kg every 3 weeks.
- Dose Escalation: DS-6157a 3.2 mg/kg: Participants with advanced GIST who received an IV infusion of DS-6157a 3.2 mg/kg every 3 weeks.
- Dose Escalation: DS-6157a 4.8 mg/kg: Participants with advanced GIST who received an IV infusion of DS-6157a 4.8 mg/kg every 3 weeks.
- Dose Escalation: DS-6157a 6.4 mg/kg: Participants with advanced GIST who received an IV infusion of DS-6157a 6.4 mg/kg every 3 weeks.
- Dose Escalation: DS-6157a 9.6 mg/kg: Participants with advanced GIST who received an IV infusion of DS-6157a 9.6 mg/kg every 3 weeks.
- Dose Escalation: DS-6157a 12.8 mg/kg: Participants with advanced GIST who received an IV infusion of DS-6157a 12.8 mg/kg every 3 weeks.
Period: Overall Study
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Started | 4 | 4 | 5 | 13 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 5 | 13 | 6 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Clinical progression | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 3 | 2 | 0
Not completed — Progressive disease | 3 | 3 | 4 | 5 | 1 | 2
Not completed — Withdrawal by patient | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 4 | 11 | 3 | 2 | 23
  >=65 years | 2 | 3 | 1 | 2 | 3 | 0 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.4) | 62.3 (17.4) | 60.8 (10.3) | 58.4 (13.0) | 55.8 (12.9) | 53.0 (9.9) | 58.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 6 | 3 | 1 | 15
  Male | 3 | 3 | 2 | 7 | 3 | 1 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 2 | 7 | 2 | 0 | 16
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 2 | 3 | 6 | 3 | 2 | 16
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 6 | 4 | 2 | 18
  Japan | 3 | 2 | 2 | 7 | 2 | 0 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Description: For hematologic toxicities, a DLT is defined as: Grade (Gr) 4 neutrophil count decreased lasting >7 days, Gr ≥3 febrile neutropenia, Gr ≥3 anemia requiring transfusion, Gr 4 anemia, Gr 4 platelet count decreased, Gr ≥3 platelet count decreased lasting >7 days or associated with clinically significant hemorrhage and/or requiring transfusion, and Gr 4 lymphocyte count decreased lasting ≥14 days. For non-hematologic, non-hepatic major organ toxicities, a DLT is all TEAEs of Gr ≥3 except: Gr 3 fatigue lasting <7 days, Gr 3 nausea, vomiting, diarrhea, or anorexia that has resolved to Gr ≤2 within 3 days with maximal medical management, Gr 3 isolated lab findings not associated with signs or symptoms including alkaline phosphatase increased, hyperuricemia, serum amylase increased, and lipase increased, and Gr 3 hyponatremia lasting <72 hours developed from Gr 1 at baseline. Symptomatic Gr 4 events were considered DLTs unless there was evidence it was associated with disease progression.
Time Frame: Cycle 1 Day 1 to Day 21 (each cycle is 21 days)
Population: Dose-limiting toxicities were assessed in the Dose Limiting Toxicity Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 3 | 5 | 11 | 6 | 2
Participants | 0 | 0 | 0 | 1 | 1 | 2

2. Primary Outcome: Number of Participants With Most Frequently Reported (≥10%) Any Grade Treatment-emergent Adverse Events (TEAEs) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Description: Treatment-emergent AEs (TEAEs) are adverse events with an onset date during the on-treatment period. Adverse events will be graded according to NCI CTCAE Version 5.0 and coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA) version 24.1.
Time Frame: Baseline up to 30 days after end of treatment, up to approximately 1 year 10 months post-treatment
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
Participants
  Any TEAE | 4 | 4 | 5 | 13 | 6 | 2
  Anemia | 3 | 2 | 4 | 6 | 3 | 1
  Febrile neutropenia | 0 | 0 | 0 | 0 | 1 | 1
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 1
  Palpitations | 0 | 0 | 0 | 0 | 0 | 1
  Sinus tachycardia | 0 | 0 | 0 | 2 | 1 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 1
  Hypothyroidism | 1 | 0 | 1 | 0 | 0 | 0
  Eye disorder | 1 | 0 | 0 | 0 | 0 | 0
  Lacrimation increased | 0 | 0 | 0 | 0 | 1 | 0
  Vitreous floaters | 0 | 1 | 0 | 0 | 0 | 0
  Abdominal distension | 0 | 1 | 1 | 1 | 0 | 1
  Abdominal pain | 1 | 2 | 1 | 2 | 1 | 2
  Abdominal pain lower | 0 | 0 | 1 | 0 | 0 | 0
  Abdominal pain upper | 1 | 0 | 0 | 0 | 0 | 0
  Anal fissure | 0 | 0 | 0 | 0 | 1 | 0
  Ascites | 0 | 0 | 1 | 0 | 0 | 0
  Constipation | 1 | 2 | 2 | 5 | 2 | 2
  Diarrhea | 0 | 0 | 1 | 3 | 1 | 1
  Dyspepsia | 0 | 1 | 0 | 0 | 1 | 1
  Flatulence | 0 | 1 | 0 | 0 | 0 | 0
  Gastritis | 1 | 0 | 0 | 0 | 0 | 0
  Gastrooesophageal reflux disease | 1 | 0 | 0 | 1 | 1 | 0
  Haematemesis | 1 | 0 | 0 | 0 | 0 | 0
  Intestinal perforation | 0 | 0 | 0 | 0 | 1 | 0
  Nausea | 3 | 3 | 3 | 11 | 6 | 2
  Upper gastrointestinal haemorrhage | 0 | 0 | 1 | 0 | 0 | 0
  Varices oesophageal | 0 | 0 | 1 | 0 | 0 | 0
  Vomiting | 1 | 2 | 2 | 4 | 1 | 2
  Asthenia | 0 | 0 | 1 | 0 | 0 | 0
  Chest discomfort | 1 | 0 | 0 | 0 | 0 | 0
  Fatigue | 3 | 1 | 3 | 6 | 2 | 2
  Influenza like illness | 1 | 0 | 0 | 0 | 0 | 0
  Injection site reaction | 0 | 1 | 0 | 0 | 0 | 0
  Malaise | 0 | 1 | 0 | 0 | 0 | 0
  Mucosal inflammation | 1 | 0 | 0 | 0 | 0 | 0
  Oedema peripheral | 1 | 1 | 3 | 1 | 0 | 2
  Pyrexia | 1 | 0 | 2 | 4 | 0 | 0
  Hepatic function abnormal | 0 | 0 | 0 | 1 | 1 | 0
  Portal hypertension | 0 | 0 | 1 | 0 | 0 | 0
  Portal vein thrombosis | 0 | 1 | 0 | 1 | 0 | 0
  Bronchitis | 0 | 0 | 1 | 0 | 0 | 0
  COVID-19 | 1 | 0 | 0 | 0 | 0 | 0
  Eye infection | 0 | 0 | 0 | 0 | 1 | 0
  Herpes zoster | 0 | 0 | 1 | 0 | 0 | 0
  Pneumonia | 0 | 0 | 0 | 0 | 0 | 1
  Upper respiratory tract infection | 0 | 1 | 0 | 0 | 0 | 0
  Contusion | 1 | 0 | 0 | 0 | 0 | 1
  Fall | 1 | 0 | 1 | 1 | 0 | 0
  Infusion related reaction | 0 | 0 | 0 | 3 | 1 | 0
  Procedural pain | 1 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 2 | 1 | 2 | 3 | 1 | 0
  Aspartate aminotransferase increased | 1 | 1 | 2 | 3 | 1 | 1
  Blood albumin decreased | 0 | 0 | 0 | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 0 | 2 | 1 | 1
  Blood creatinine increased | 0 | 0 | 0 | 1 | 2 | 0
  Blood potassium decreased | 0 | 0 | 0 | 0 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 1 | 1 | 1 | 1
  Neutrophil count decreased | 0 | 0 | 0 | 5 | 4 | 0
  Platelet count decreased | 0 | 1 | 2 | 4 | 5 | 1
  Protein total decreased | 0 | 0 | 0 | 0 | 0 | 1
  Weight decreased | 0 | 0 | 1 | 2 | 0 | 1
  White blood cell count decreased | 0 | 0 | 0 | 3 | 5 | 1
  Decreased appetite | 3 | 2 | 4 | 6 | 4 | 2
  Dehydration | 1 | 0 | 0 | 1 | 1 | 2
  Hyperglycaemia | 0 | 1 | 1 | 1 | 0 | 0
  Hyperkalaemia | 1 | 0 | 1 | 0 | 0 | 0
  Hyperphosphataemia | 0 | 0 | 1 | 0 | 0 | 0
  Hyperuricaemia | 0 | 1 | 1 | 1 | 2 | 0
  Hypoalbuminaemia | 0 | 1 | 2 | 2 | 0 | 0
  Hypocalcaemia | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycaemia | 1 | 0 | 0 | 1 | 0 | 0
  Hypokalaemia | 0 | 1 | 1 | 2 | 1 | 1
  Hyponatraemia | 1 | 1 | 0 | 0 | 0 | 1
  Hypophosphataemia | 0 | 1 | 0 | 1 | 0 | 0
  Athralgia | 1 | 0 | 1 | 0 | 0 | 0
  Arthritis | 1 | 0 | 0 | 0 | 0 | 0
  Back pain | 1 | 0 | 0 | 0 | 2 | 0
  Flank pain | 0 | 0 | 1 | 0 | 0 | 0
  Muscle fatigue | 0 | 1 | 0 | 0 | 0 | 0
  Muscle spasms | 0 | 1 | 0 | 0 | 0 | 0
  Muscular weakness | 0 | 0 | 0 | 1 | 1 | 0
  Myalgia | 1 | 1 | 0 | 0 | 0 | 0
  Disturbance in attention | 0 | 0 | 0 | 0 | 1 | 0
  Dizziness | 1 | 0 | 0 | 4 | 1 | 2
  Dysarthria | 0 | 0 | 0 | 0 | 1 | 0
  Dysgeusia | 0 | 1 | 1 | 2 | 0 | 0
  Headache | 1 | 1 | 1 | 4 | 0 | 0
  Hyperaesthesia | 0 | 0 | 1 | 0 | 1 | 0
  Peripheral sensory neuropathy | 0 | 0 | 0 | 0 | 1 | 0
  Taste disorder | 1 | 0 | 0 | 0 | 0 | 0
  Anxiety | 0 | 0 | 1 | 1 | 0 | 1
  Confusional state | 0 | 0 | 0 | 0 | 1 | 1
  Delirium | 0 | 0 | 0 | 0 | 0 | 1
  Insomnia | 1 | 2 | 1 | 2 | 2 | 0
  Haematuria | 0 | 1 | 0 | 0 | 0 | 0
  Pollakiuria | 0 | 0 | 1 | 1 | 0 | 0
  Proteinuria | 1 | 0 | 0 | 1 | 1 | 0
  Renal disorder | 0 | 0 | 0 | 0 | 1 | 0
  Urinary tract obstruction | 0 | 0 | 0 | 0 | 0 | 1
  Pelvic pain | 0 | 0 | 0 | 0 | 1 | 0
  Cough | 1 | 0 | 0 | 3 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 3 | 2 | 0
  Dyspnoea exertional | 0 | 2 | 0 | 1 | 0 | 0
  Epistaxis | 1 | 0 | 0 | 0 | 1 | 0
  Hiccups | 0 | 0 | 1 | 0 | 0 | 1
  Pulmonary embolism | 0 | 0 | 0 | 0 | 0 | 1
  Rhinorrhoea | 0 | 0 | 1 | 0 | 0 | 0
  Sleep apnoea syndrome | 0 | 0 | 0 | 0 | 0 | 1
  Alopecia | 0 | 0 | 1 | 0 | 1 | 0
  Dry skin | 1 | 2 | 3 | 0 | 0 | 1
  Hyperhidrosis | 1 | 0 | 1 | 1 | 1 | 0
  Rash maculo-papular | 1 | 1 | 1 | 0 | 2 | 0
  Rash papular | 1 | 0 | 0 | 0 | 0 | 0
  Skin fissures | 0 | 0 | 0 | 0 | 1 | 0
  Deep vein thrombosis | 0 | 0 | 0 | 0 | 0 | 2
  Hot flush | 0 | 1 | 0 | 0 | 0 | 0
  Hypertension | 1 | 1 | 0 | 2 | 0 | 1
  Hypotension | 0 | 0 | 0 | 2 | 0 | 1

3. Primary Outcome: Objective Response Rate (ORR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Expansion)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Duration of Response (DoR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Expansion)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Expansion: Cohort 1 (3rd Line or Later) Treated at RDE | Dose Expansion: Cohort 2 (2nd Line) Treated at RDE
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Disease Control Rate (DCR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Expansion)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Expansion: Cohort 1 (3rd Line or Later) Treated at RDE | Dose Expansion: Cohort 2 (2nd Line) Treated at RDE
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Progression-free Survival (PFS) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Expansion)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Expansion: Cohort 1 (3rd Line or Later) Treated at RDE | Dose Expansion: Cohort 2 (2nd Line) Treated at RDE
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Plasma Concentration-time Curve up to the Last Quantifiable Time (AUClast) for DS-6157a and Total Anti-GPR20 Antibody Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: Cycle 1, Day 1: Predose, postdose, and 2 hours (hr), 4 hr, 7 hr postdose to Cycle 8, Day 1 predose (each cycle is 21 days)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
day*ug/mL
  DS-6157a: Cycle 1 | 181 (18.2) | 399 (178) | 574 (150) | 776 (346) | 1530 (507) | 2140 (351)
  DS-6157a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  DS-6157a: Cycle 3 | 223 (76.6) | 761 (47.3) | 733 (425) | 1520 (654) | 2570 (11.9) |
  Total anti-GPR20 antibody: Cycle 1 | 176 (22.6) | 425 (203) | 549 (111) | 730 (349) | 1530 (495) | 1980 (256)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 218 (76.9) | 731 (40.4) | 676 (428) | 1570 (746) | 2450 (217) |

8. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Plasma Concentration-time Curve up to the Last Quantifiable Time (AUClast) for MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
day*ng/mL
  MAAA-1181a: Cycle 1 | 6.85 (2.16) | 19 (2.49) | 20.5 (5.53) | 51.8 (23.8) | 74.8 (30.2) | 111 (27.9)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  MAAA-1181a: Cycle 3 | 5.95 (0.94) | 22.3 (3.58) | 22.8 (10.4) | 75.9 (55.9) | 70.6 (30.4) |

9. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Plasma Concentration-time Curve in the Dosing Interval (AUCtau) for DS-6157a and Total Anti-GPR20 Antibody Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 12 | 6 | 2
day*ug/mL
  DS-6157a: Cycle 1: number analyzed (Participants) | 4 | 4 | 4 | 12 | 6 | 2
  DS-6157a: Cycle 1 | 181 (18.3) | 400 (157) | 512 (67.1) | 821 (371) | 1570 (401) | 1690 (499)
  DS-6157a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  DS-6157a: Cycle 3 | 250 (36.8) | 718 (35.1) | 780 (342) | 1430 (458) | 2400 (240) |
  Total anti-GPR20 antibody: Cycle 1 | 176 (22.8) | 427 (182) | 549 (113) | 781 (363) | 1570 (394) | 1590 (388)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 251 (31.1) | 691 (24.6) | 733 (344) | 1460 (538) | 2270 (60.8) |

10. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Plasma Concentration-time Curve in the Dosing Interval (AUCtau) for MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 12 | 5 | 2
day*ng/mL
  MAAA-1181a: Cycle 1 | 6.85 (2.16) | 19.7 (4.01) | 20.4 (5.55) | 49.5 (23.5) | 69.1 (30.7) | 98.5 (18.5)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 0
  MAAA-1181a: Cycle 3 | 6.48 (0.52) | 21.8 (3.86) | 27.6 (5.07) | 70.7 (61.1) | 66.9 (25) |

11. Secondary Outcome: Pharmacokinetic Analysis: Time to Maximum Plasma Concentration (Tmax) for DS-6157a, Total Anti-GPR20 Antibody, and MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
hours
  DS-6157a: Cycle 1 | 2.59 (1.04) | 2.09 (0.83) | 2.75 (1.53) | 2.71 (1.54) | 2.86 (2.82) | 2.7 (1.52)
  DS-6157a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  DS-6157a: Cycle 3 | 1.24 (0.99) | 3.75 (1.23) | 2.07 (1.65) | 2.58 (2.48) | 4.05 (4.71) |
  Total anti-GPR20 antibody: Cycle 1 | 2.17 (0.96) | 3.06 (1.84) | 2.36 (0.83) | 2.53 (1.26) | 2.62 (0.99) | 1.77 (0.21)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 1.81 (1.02) | 4.24 (3.45) | 2.07 (1.65) | 4.96 (7.82) | 2.47 (0.12) |
  MAAA-1181a: Cycle 1 | 10.5 (8.36) | 7.26 (2.62) | 11.1 (8.96) | 8.42 (7.16) | 34.17 (65.53) | 3.76 (0.01)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  MAAA-1181a: Cycle 3 | 11.52 (9.85) | 18.61 (23.73) | 10.59 (8.32) | 19.63 (13.53) | 15.72 (11.79) |

12. Secondary Outcome: Pharmacokinetic Analysis: Maximum Plasma Concentration (Cmax) for DS-6157a and Total Anti-GPR20 Antibody Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
ug/mL
  DS-6157a: Cycle 1 | 32.3 (4.01) | 71.4 (15.7) | 100 (6.1) | 142 (28.7) | 227 (33.7) | 291 (88.4)
  DS-6157a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  DS-6157a: Cycle 3 | 37 (0.55) | 90.8 (13.8) | 118 (16.8) | 162 (51.9) | 280 (47.4) |
  Total anti-GPR20 antibody: Cycle 1 | 32.3 (1.89) | 78.8 (23.3) | 98.6 (7.62) | 137 (33.7) | 237 (26.2) | 279 (61.5)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 35.2 (2.38) | 89.9 (15.1) | 111 (12.4) | 160 (42.9) | 267 (48.1) |

13. Secondary Outcome: Pharmacokinetic Analysis: Maximum Plasma Concentration (Cmax) for MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
ng/mL
  MAAA-1181a: Cycle 1 | 1.5 (0.88) | 4.51 (2.03) | 4 (1.19) | 12.8 (11.4) | 14.6 (3.36) | 19.4 (1.2)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  MAAA-1181a: Cycle 3 | 1.12 (0.25) | 3.48 (1.18) | 4.78 (1.35) | 9.76 (5.13) | 7.92 (1.4) |

14. Secondary Outcome: Pharmacokinetic Analysis: Lowest Concentration Reached After a Single Dose (Ctrough) for DS-6157a and Total Anti-GPR20 Antibody Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 3 | 5 | 10 | 5 | 2
ug/mL
  DS-6157a: Cycle 1 | 3.09 (0.57) | 9.1 (2.16) | 13.9 (12.9) | 15.8 (9.27) | 27.9 (13.6) | 7.16 (6)
  DS-6157a: Cycle 3: number analyzed (Participants) | 2 | 3 | 3 | 6 | 2 | 0
  DS-6157a: Cycle 3 | 5.1 (1.87) | 14.7 (1.68) | 21 (8.6) | 28.6 (7.21) | 52.8 (12) |
  Total anti-GPR20 antibody: Cycle 1 | 3.54 (0.84) | 8.96 (0.36) | 8.93 (4.9) | 14.3 (10.1) | 24.3 (12.6) | 6.45 (4.82)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 2 | 3 | 3 | 6 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 6.32 (0.87) | 11.7 (6.05) | 23 (9.76) | 30 (10) | 58.8 (13.2) |

15. Secondary Outcome: Pharmacokinetic Analysis: Lowest Concentration Reached After a Single Dose (Ctrough) for MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 3 | 5 | 10 | 5 | 2
ng/mL
  MAAA-1181a: Cycle 1 | 0.05 (0.01) | 0.13 (0.03) | 0.17 (0.10) | 0.41 (0.35) | 0.54 (0.28) | 0.16 (0.20)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 2 | 3 | 3 | 6 | 2 | 0
  MAAA-1181a: Cycle 3 | 0.07 (0.01) | 0.18 (0.03) | 0.37 (0.21) | 1.16 (1.4) | 0.65 (0.27) |

16. Secondary Outcome: Pharmacokinetic Analysis: Terminal Elimination Half-life (t1/2) for DS-6157a, Total Anti-GPR20 Antibody, and MAAA-1181a Following Intravenous Administration of DS-6157a
Description: The plasma PK parameters were estimated using standard noncompartmental methods.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 12 | 6 | 2
day
  DS-6157a: Cycle 1: number analyzed (Participants) | 4 | 4 | 4 | 12 | 6 | 2
  DS-6157a: Cycle 1 | 9.05 (1.02) | 8.37 (4.91) | 9.73 (3.27) | 10 (4.61) | 7.58 (2.01) | 2.7 (1.52)
  DS-6157a: Cycle 3: number analyzed (Participants) | 3 | 3 | 4 | 7 | 2 | 0
  DS-6157a: Cycle 3 | 9.1 (5.38) | 12.8 (4) | 9.61 (5.52) | 14.7 (2.64) | 11.2 (3.95) |
  Total anti-GPR20 antibody: Cycle 1 | 9.35 (2.08) | 8.49 (3.61) | 9.47 (3.45) | 9.69 (4.5) | 7.94 (2.73) | 11.8 (4.72)
  Total anti-GPR20 antibody: Cycle 3: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 0
  Total anti-GPR20 antibody: Cycle 3 | 10.7 (3.49) | 10 (4.24) | 13.2 (9.28) | 14.4 (1.66) | 12.7 (4.03) |
  MAAA-1181a: Cycle 1: number analyzed (Participants) | 4 | 4 | 5 | 12 | 5 | 2
  MAAA-1181a: Cycle 1 | 5.05 (1.23) | 4.29 (1.29) | 5.35 (1.39) | 6.52 (3.59) | 4.73 (0.59) | 7.27 (2.77)
  MAAA-1181a: Cycle 3: number analyzed (Participants) | 3 | 3 | 3 | 5 | 2 | 0
  MAAA-1181a: Cycle 3 | 5.45 (1.8) | 5.67 (1.06) | 6.37 (1.32) | 7.72 (1.71) | 6.67 (1.98) |

17. Secondary Outcome: Best Overall Response Rate Following Intravenous Administration of DS-6157a in Participants With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Escalation)
Description: Based on Response Evaluation Criteria In Solid Tumors guidelines, complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions).
Time Frame: Baseline up to long-term follow up (defined as until the start of a new anti-cancer treatment, PD, death, lost to follow up, withdrawal of consent, or at the discretion of the Investigator, whichever occurs first), up to approximately 1 year 10 months.
Population: Best overall response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 13 | 6 | 2
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 1 | 0 | 0
  Stable disease (SD) | 2 | 3 | 3 | 7 | 2 | 0
  Progressive disease (PD) | 2 | 0 | 2 | 3 | 1 | 2
  Not evaluable (NE) | 0 | 1 | 0 | 2 | 3 | 0

18. Secondary Outcome: Progression-free Survival (PFS) Following Intravenous Administration of DS-6157a in Participants With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Escalation)
Description: Progression-free survival (PFS) is defined as the time from randomization/start of study treatment to the date of event defined as the first documented radiological progression or death due to any cause.
Time Frame: Baseline up to the date of the first documented radiological progression or death due to any cause, whichever occurs first, up to approximately 1 year 10 months
Population: Progression-free survival was assessed in participants with available data (events) in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 4 | 3 | 4 | 7 | 3 | 2
months | 2.6 [1.2 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis. | 6.9 [5.1 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis. | 10.4 [0.9 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis. | 4.2 [0.8 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis. | 3.6 [1.2 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis. | 1.5 [1.3 to NA] — The maximum 95% confidence interval limit could not be estimated due to insufficient number of events for analysis.

19. Secondary Outcome: Objective Response Rate (ORR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Escalation)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Duration of Response (DoR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Escalation)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Disease Control Rate (DCR) Following Intravenous Administration of DS-6157a in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) (Dose Escalation)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Anti-drug Antibodies Against DS-6157a Following Intravenous Administration of DS-6157a in Participants With Advanced Gastrointestinal Stromal Tumors (GIST)
Time Frame: Baseline up to 5 years post-treatment
Population: This outcome measure was not assessed due to early study termination.
Arm/Group | Dose Expansion: Cohort 1 (3rd Line or Later) Treated at RDE | Dose Expansion: Cohort 2 (2nd Line) Treated at RDE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 30 days after last administration of study drug, up to approximately 1 year 10 months.
Description: An adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. AEs were graded according to NCI CTCAE Version 5.0. AEs are only reported for the Dose Escalation phase. The Dose Expansion phase was not conducted since the study terminated early.
Arm/Group | Dose Escalation: DS-6157a 1.6 mg/kg | Dose Escalation: DS-6157a 3.2 mg/kg | Dose Escalation: DS-6157a 4.8 mg/kg | Dose Escalation: DS-6157a 6.4 mg/kg | Dose Escalation: DS-6157a 9.6 mg/kg | Dose Escalation: DS-6157a 12.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/4 | 2/5 | 2/13 | 1/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 1/5 | 2/13 | 3/6 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 13/13 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: DS-6157a 1.6 mg/kg (N=4) | Dose Escalation: DS-6157a 3.2 mg/kg (N=4) | Dose Escalation: DS-6157a 4.8 mg/kg (N=5) | Dose Escalation: DS-6157a 6.4 mg/kg (N=13) | Dose Escalation: DS-6157a 9.6 mg/kg (N=6) | Dose Escalation: DS-6157a 12.8 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: DS-6157a 1.6 mg/kg (N=4) | Dose Escalation: DS-6157a 3.2 mg/kg (N=4) | Dose Escalation: DS-6157a 4.8 mg/kg (N=5) | Dose Escalation: DS-6157a 6.4 mg/kg (N=13) | Dose Escalation: DS-6157a 9.6 mg/kg (N=6) | Dose Escalation: DS-6157a 12.8 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 4 | 6 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 5 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 11 | 6 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 4 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 3 | 6 | 2 | 2
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 3 | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 2 | 4 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 2 | 3 | 1 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 3 | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 5 | 4 | 0
Platelet count decreased (Investigations) | 0 | 1 | 2 | 4 | 5 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 3 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 4 | 6 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 4 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 4 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04276415/Prot_SAP_000.pdf